CLINICAL TRIAL: NCT00779558
Title: Heparin and Catheter-related Thrombosis in Neonates and Infants Following Cardiac Surgery
Brief Title: Heparin and the Reduction of Thrombosis (HART) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alan Schroeder, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-11132007-879
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study drug (Active Comparator): Heparin sulfate infusion at 10 units/kg/hour
  Interventions: Drug: Heparin sulfate infusion at 10 units/kg/hour
- Placebo (Placebo Comparator): Placebo - normal saline infusion
  Interventions: Drug: Placebo infusion

INTERVENTIONS:
Drug: Heparin sulfate infusion at 10 units/kg/hour — Infusion of heparin to prevent central line thrombosis in infants after cardiac surgery
  Other Names: heparin
  Arms: Study drug
Drug: Placebo infusion — Infusion of normal saline
  Arms: Placebo

SUMMARY:
Heparin is frequently used in central venous catheters (CVCs) in post-operative cardiac patients. It remains unclear if a heparin infusion, compared to a normal saline infusion, prevents thrombosis of CVCs after surgery. This study will answer the question: does a low-dose heparin infusion (10 units/kg/h) prevent thrombosis, compared to a normal saline infusion, in patients less than one year of age after cardiac surgery?

DETAILED DESCRIPTION:
Patients are contacted pre-operatively and their parents consented. The following criteria apply:

Inclusion criteria:

All infants < 1 year of age undergoing cardiac surgery at Lucile Packard Children's Hospital

Exclusion Criteria:

Known coagulopathy History of clinically significant bleeding (GI, cranial, pulmonary) Need for therapeutic heparinization ECMO

Randomization and blinding are performed in the Pharmacy. The intervention is initiated at the intensive care unit physician's discretion, generally within the 1st 24 hours post-operatively. The study is terminated when all catheters have been discontinued or at POD #14, whichever occurs first.

Thrombosis is demonstrated by echocardiogram or ultrasound performed at

1 - 3 days, 5 - 7 days, and 10 - 14 days after initiation of the study drug.

The following are calculations for statistical analysis:

Sample size determination - Using 2 - sided alpha = 0.05 and Beta = 0.2, and assuming a baseline thrombosis incidence of 20%, 160 patients are required to detect an effect size of 15%.

ELIGIBILITY:
Inclusion Criteria:

* All infants < 1 year of age undergoing cardiac surgery at Lucile Packard Children's Hospital & #xA

Exclusion Criteria:

* Known coagulopathy
* History of clinically significant bleeding (GI, cranial, pulmonary)
* Need for therapeutic heparinization
* ECMO

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Roth M.D., M.P.H., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Schroeder AR, Axelrod DM, Silverman NH, Rubesova E, Merkel E, Roth SJ. A continuous heparin infusion does not prevent catheter-related thrombosis in infants after cardiac surgery. Pediatr Crit Care Med. 2010 Jul;11(4):489-95. doi: 10.1097/PCC.0b013e3181ce6e29. PMID 20101197

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Drug | Placebo
Started | 57 | 44
Completed | 53 | 37
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug | Placebo | Total
Number analyzed (Participants) | 53 | 37 | 90
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.1 (2.7) | 4.3 (3.2) | 4.2 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 14 | 38
  Male | 29 | 23 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 43 | 31 | 74
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Thrombosis
Description: Echocardiographic evidence of thrombosis while on study drug
Time Frame: While on study drug, which was continued until all catheters were removed, or 2 weeks (whichever came first). Echoes were performed after 24-48 hours and then every 3-5 days
Measure: Number; unit: participants
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 53 | 37
participants | 8 | 6

2. Secondary Outcome: Total PRBCs Transfused
Time Frame: While on study drug, which was continued until all catheters were removed, or 2 weeks (whichever came first)
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 53 | 37
mL/kg | 8.8 (13) | 5.6 (10.6)

3. Secondary Outcome: Days to Extubation
Time Frame: While on study drug, which was continued until all catheters were removed, or 2 weeks (whichever came first)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 53 | 37
days | 3.5 (3.7) | 3.3 (3.1)

4. Secondary Outcome: Cardiac ICU Length of Stay
Time Frame: While on study drug, which was continued until all catheters were removed, or 2 weeks (whichever came first)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 53 | 37
days | 10 (9.7) | 6.9 (4.7)

5. Secondary Outcome: Need for Antibiotics
Time Frame: While on study drug, which was continued until all catheters were removed, or 2 weeks (whichever came first)
Measure: Number; unit: participants
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 53 | 37
participants | 14 | 9

ADVERSE EVENTS:
Arm/Group | Study Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/37
Other Adverse Events (participants affected / at risk) | 0/53 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes